CLINICAL TRIAL: NCT05392855
Title: Symptom Based Performance of Airway Clearance Therapy After Starting Highly Effective CFTR Modulator Therapy for Cystic Fibrosis
Brief Title: Symptom Based Performance of Airway Clearance After Starting Highly Effective Modulators for Cystic Fibrosis (SPACE-CF)
Acronym: SPACE-CF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment, low interest from participant population
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Zach Holliday, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2088922
Record Dates: First submitted 2022-05-20; First posted 2022-05-26 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Cystic Fibrosis; Mucociliary Clearance Defect
Keywords: Cystic Fibrosis; Mucociliary clearance; Highly Effective CFTR Modulator Therapy
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial design with 2:1 randomization (2 to symptom driven to 1 in continuous) for this pilot study to determine if intermittent and symptom-driven airway clearance after starting Elexacaftor-Tezacaftor-Ivacaftor (ETI) therapy can be determined to be non-inferior to continuing airway clearance therapies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Symptom driven (Experimental): Symptom driven performance of airway clearance regimen
  Interventions: Other: Symptom driven performance of airway clearance
- Continuous (Active Comparator): Continuous performance of baseline daily airway clearance regimen
  Interventions: Other: Continuous daily performance of airway clearance

INTERVENTIONS:
Other: Symptom driven performance of airway clearance — Perform symptom driven/intermittent airway clearance therapy with frequency based off of patient's daily symptoms including mobilization therapy (high-frequency chest compression or vest device, intrapulmonary percussive ventilator, positive expiratory pressure device) and inhaled/nebulized therapies of albuterol, hypertonic saline and dornase alfa for the 12 week study period.
  Arms: Symptom driven
Other: Continuous daily performance of airway clearance — Continue run-in protocol of twice daily airway clearance using twice daily mobilization therapy (high-frequency chest compression or vest device, intrapulmonary percussive ventilator, positive expiratory pressure device) and inhaled/nebulized therapies of albuterol, hypertonic saline and dornase alfa for the 12 week study period.
  Arms: Continuous

SUMMARY:
Cystic Fibrosis (CF) is an autosomal recessive disease cause by a mutation in the cystic fibrosis transmembrane conductance regulator (CFTR) manifesting in multiple organs, the most common cause of morbidity and mortality continues to be the pulmonary manifestation. CFTR dysfunction leads to reduced mucociliary clearance, impaired innate immune system function in the lungs (within the airway surface liquid [ASL] lining the epithelial barrier of the lungs) and reduced ASL hydration (stickier mucus). To try and help correct this underlying defect patients have been performing airway clearance for decades using different techniques (Percussion and postural drainage [P&PD], Positive expiratory pressure [PEP], Oscillatory positive expiratory pressure [OPEP], High-frequency chest compression [HFCC], exercise), inhaled mucolytics (Hypertonic Saline, Pulmozyme) and inhaled antibiotics. However, performing daily airway clearance can be a large burden on patients and their families with a median number of daily therapies around 7 and average time spent on therapies at almost 2 hours daily. This high treatment burden leads many patients to have reduced adherence to their regimens and multiple studies have shown around 20% of patients performing no daily airway clearance. Since the release of highly effective CFTR modulator therapy patients have experienced improvements in lung function measurements and imaging-based ventilation measurements, reduction in pulmonary exacerbations, and improvement in daily symptom scores. Over 80% of patients and their families and over 95% of clinicians in the United States support the idea of trials looking into the simplification of airway clearance regimens. Combining the inability of most patients to complete their daily regimens, patient and clinician interest in treatment simplification research, and the overwhelming cost of most inhaled medications in cystic fibrosis with the improvement in mucociliary transport and symptoms with highly effective modulator therapy suggests a research program aimed at reducing the treatment burden of daily airway clearance should be considered. The investigators propose the following: determine if there is additional benefit in continuous airway clearance regimens after starting Elexacaftor-Tezacaftor-Ivacaftor (ETI) and if so, is this benefit noticeable on pulmonary function testing and imaging.

DETAILED DESCRIPTION:
This will be a randomized controlled trial design with 2:1 randomization (2 to symptom driven to 1 in continuous) for this pilot study to determine if symptom-driven airway clearance after starting Elexacaftor-Tezacaftor-Ivacaftor (ETI) therapy is feasible and can eventually determine if it is non-inferior to continuing airway clearance therapies. The study will be performed as an intention to treat protocol. All participants who are eligible and enrolled will be asked to perform airway clearance twice daily for 12 weeks prior to randomization and then will be followed for 12 weeks including study visits at week 0, week 4, week 8, and week 12. The study will require no change in current use of inhaled antibiotics nor adjust the frequency of the medication during the study. Airway clearance methods to be recorded include aerobika or flutter valve, high frequency chest oscillation therapy (vest), intrapulmonary percussive ventilator, or exercise performed specially for airway clearance. The medications to be monitored included nebulized Albuterol, nebulized hypertonic saline, nebulized Pulmozyme, and nebulized mannitol. The continuous arm (control arm) will be asked to perform airway clearance twice daily for the entirety of the study and record all therapies performed daily. The symptom driven arm will perform airway clearance on their own discretion, whether this be from steady decline in baseline respiratory status or acute flair of symptoms related to infectious etiology. At baseline participants will undergo pulmonary function testing, sputum/throat culture and Cystic Fibrosis Questionnaire Revise (CFQ-R). On week 0, week 4, week 8 and week 12 visits the participants will undergo pulmonary function testing and CFQ-R with addition of sputum/throat cultures on week 12. Between each study visit participants will be asked to perform home spirometry once weekly for the 12-week trial period. For participants enrolled in the continuous group the investigators will ask for participants to perform home spirometry after either twice daily airway clearance routine or for the symptom-based group to perform at roughly the same time of day for each test. Participants will also be asked to keep a daily cystic fibrosis diary during the run-in period and study period in which participants will record if, and how frequent, participants use any airway clearance medications or devices during the day. A reduction in percent predicted forced expiratory volume in 1 second (ppFEV1%) or percent predicted forced vital capacity (ppFVC%) of more than 10% in laboratory PFT testing for 2 consecutive weeks will be deemed an adverse event and lead to the participant in the symptom driven arm being instructed to perform daily airway clearance therapy. A reduction in ppFEV1% and/or ppFVC% in home spirometry by more than 10% will trigger a need for in lab PFT testing to determine if participants have developed an adverse event leading to performing daily airway clearance therapy or if participants are to continue symptom-based airway clearance. Other criteria for participants to be evaluate in-person between study visits include use of daily airway clearance for more than 7 consecutive days in the symptom-based arm or signs and symptoms of a possible acute pulmonary exacerbation. If participants develop an exacerbation from an identifiable cause other than their primary CF lung disease (viral infection, asthma exacerbation, pulmonary embolism, etc.) participants will undergo appropriate treatment, and while the event will be deemed an adverse event, participants will continue with their current treatment protocol. Participants who are treated for an acute severe pulmonary exacerbation requiring IV antibiotics and/or hospitalization will either continue in the continuous treatment arm or if in the symptom driven arm be instructed to perform daily airway clearance for the duration of the study. In participants with concurrent asthma diagnoses, the investigators will not require any discontinuation of additional inhaler/nebulized therapies that are asthma specific, but no bronchodilators will be started specifically for the study.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years at the time of recruitment
* treatment with Elexacaftor-Tezacaftor-Ivacaftor for > 90 days prior to enrollment
* willing to continue twice daily airway clearance for a minimum of 90 days and up to180 days if enrolled in the continuing treatment arm
* no exacerbations in the last 28 days

Exclusion Criteria:

* active smoking or vaping (tobacco, marijuana, recreational drugs)
* recent change in chronic airway clearance regimen with the last 28 days
* inability to tolerate airway clearance or intolerance to either/or hypertonic saline and Pulmozyme
* current treatment for an acute pulmonary exacerbation
* ongoing therapy for Nontuberculous Mycobacterium (NTM)
* investigational drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Absolute change in percent predicted FEV1 (ppFEV1) from week 0 to week 12 in symptom driven airway clearance arm | 12 weeks
  Difference between symptom driven airway clearance arm and continue daily airway clearance arm in the absolute change in ppFEV1 from Week 0 to Week 12
Absolute change in percent predicted FVC (ppFVC) from week 0 to week 12 in symptom driven airway clearance arm | 12 weeks
  Difference between symptom driven airway clearance arm and continue daily airway clearance arm in the absolute change in ppFVC from Week 0 to Week 12

SECONDARY OUTCOMES:
Absolute change in respiratory symptoms based upon Cystic Fibrosis Questionnaire Revise score | 12 weeks
  Difference between symptom driven airway clearance arm and continue daily airway clearance arm in the absolute change in respiratory symptoms based upon Cystic Fibrosis Questionnaire Revise score (CFQ-R). Scores for the CFQ-R range from 0-100 with higher scores analogous to better outcomes.
Incidence of adverse events (AE) in the symptom driven airway clearance arm | 12 weeks
  Difference between symptom driven airway clearance arm and continue daily airway clearance arm in the proportion of participants with at least one event per week
Frequency of performance of airway clearance in symptom driven airway clearance arm | 12 weeks
  Difference between symptom driven airway clearance arm and continue daily airway clearance arm in the absolute difference of performance of airway clearance
Change in airway colonization with S. aureus or P. aeruginosa | 12 weeks
  Difference between symptom based airway clearance arm and continue daily airway clearance arm in the absolute difference in sputum/throat cultures positive for S. aureus or P. aeruginosa

CONTACTS AND LOCATIONS:
Overall Officials: Zach Holliday, MD, Principal Investigator — University of Missouri School of Medicine
Locations (1):
- University of Missouri Hospital and Clinics, Columbia, Missouri, United States

REFERENCES:
- [Background] Elborn JS. Cystic fibrosis. Lancet. 2016 Nov 19;388(10059):2519-2531. doi: 10.1016/S0140-6736(16)00576-6. Epub 2016 Apr 29. PMID 27140670
- [Background] Henderson AG, Ehre C, Button B, Abdullah LH, Cai LH, Leigh MW, DeMaria GC, Matsui H, Donaldson SH, Davis CW, Sheehan JK, Boucher RC, Kesimer M. Cystic fibrosis airway secretions exhibit mucin hyperconcentration and increased osmotic pressure. J Clin Invest. 2014 Jul;124(7):3047-60. doi: 10.1172/JCI73469. Epub 2014 Jun 2. PMID 24892808
- [Background] Button B, Cai LH, Ehre C, Kesimer M, Hill DB, Sheehan JK, Boucher RC, Rubinstein M. A periciliary brush promotes the lung health by separating the mucus layer from airway epithelia. Science. 2012 Aug 24;337(6097):937-41. doi: 10.1126/science.1223012. PMID 22923574
- [Background] Collawn JF, Matalon S. CFTR and lung homeostasis. Am J Physiol Lung Cell Mol Physiol. 2014 Dec 15;307(12):L917-23. doi: 10.1152/ajplung.00326.2014. Epub 2014 Nov 7. PMID 25381027
- [Background] Quinton PM. Cystic fibrosis: impaired bicarbonate secretion and mucoviscidosis. Lancet. 2008 Aug 2;372(9636):415-7. doi: 10.1016/S0140-6736(08)61162-9. PMID 18675692
- [Background] Hoegger MJ, Fischer AJ, McMenimen JD, Ostedgaard LS, Tucker AJ, Awadalla MA, Moninger TO, Michalski AS, Hoffman EA, Zabner J, Stoltz DA, Welsh MJ. Impaired mucus detachment disrupts mucociliary transport in a piglet model of cystic fibrosis. Science. 2014 Aug 15;345(6198):818-22. doi: 10.1126/science.1255825. PMID 25124441
- [Background] Flume PA, Robinson KA, O'Sullivan BP, Finder JD, Vender RL, Willey-Courand DB, White TB, Marshall BC; Clinical Practice Guidelines for Pulmonary Therapies Committee. Cystic fibrosis pulmonary guidelines: airway clearance therapies. Respir Care. 2009 Apr;54(4):522-37. PMID 19327189
- [Background] Desmond KJ, Schwenk WF, Thomas E, Beaudry PH, Coates AL. Immediate and long-term effects of chest physiotherapy in patients with cystic fibrosis. J Pediatr. 1983 Oct;103(4):538-42. doi: 10.1016/s0022-3476(83)80579-4. PMID 6620013
- [Background] Mogayzel PJ Jr, Naureckas ET, Robinson KA, Mueller G, Hadjiliadis D, Hoag JB, Lubsch L, Hazle L, Sabadosa K, Marshall B; Pulmonary Clinical Practice Guidelines Committee. Cystic fibrosis pulmonary guidelines. Chronic medications for maintenance of lung health. Am J Respir Crit Care Med. 2013 Apr 1;187(7):680-9. doi: 10.1164/rccm.201207-1160oe. PMID 23540878
- [Background] Sawicki GS, Sellers DE, Robinson WM. High treatment burden in adults with cystic fibrosis: challenges to disease self-management. J Cyst Fibros. 2009 Mar;8(2):91-6. doi: 10.1016/j.jcf.2008.09.007. Epub 2008 Oct 26. PMID 18952504
- [Background] White D, Stiller K, Haensel N. Adherence of adult cystic fibrosis patients with airway clearance and exercise regimens. J Cyst Fibros. 2007 May;6(3):163-70. doi: 10.1016/j.jcf.2006.06.006. Epub 2006 Aug 10. PMID 16904388
- [Background] Ramsey BW, Davies J, McElvaney NG, Tullis E, Bell SC, Drevinek P, Griese M, McKone EF, Wainwright CE, Konstan MW, Moss R, Ratjen F, Sermet-Gaudelus I, Rowe SM, Dong Q, Rodriguez S, Yen K, Ordonez C, Elborn JS; VX08-770-102 Study Group. A CFTR potentiator in patients with cystic fibrosis and the G551D mutation. N Engl J Med. 2011 Nov 3;365(18):1663-72. doi: 10.1056/NEJMoa1105185. PMID 22047557
- [Background] Altes TA, Johnson M, Fidler M, Botfield M, Tustison NJ, Leiva-Salinas C, de Lange EE, Froh D, Mugler JP 3rd. Use of hyperpolarized helium-3 MRI to assess response to ivacaftor treatment in patients with cystic fibrosis. J Cyst Fibros. 2017 Mar;16(2):267-274. doi: 10.1016/j.jcf.2016.12.004. Epub 2017 Jan 26. PMID 28132845
- [Background] Mentore K, Froh DK, de Lange EE, Brookeman JR, Paget-Brown AO, Altes TA. Hyperpolarized HHe 3 MRI of the lung in cystic fibrosis: assessment at baseline and after bronchodilator and airway clearance treatment. Acad Radiol. 2005 Nov;12(11):1423-9. doi: 10.1016/j.acra.2005.07.008. PMID 16253854
- [Background] McMahon CJ, Dodd JD, Hill C, Woodhouse N, Wild JM, Fichele S, Gallagher CG, Skehan SJ, van Beek EJ, Masterson JB. Hyperpolarized 3helium magnetic resonance ventilation imaging of the lung in cystic fibrosis: comparison with high resolution CT and spirometry. Eur Radiol. 2006 Nov;16(11):2483-90. doi: 10.1007/s00330-006-0311-5. Epub 2006 Jul 27. PMID 16871384
- [Background] Middleton PG, Mall MA, Drevinek P, Lands LC, McKone EF, Polineni D, Ramsey BW, Taylor-Cousar JL, Tullis E, Vermeulen F, Marigowda G, McKee CM, Moskowitz SM, Nair N, Savage J, Simard C, Tian S, Waltz D, Xuan F, Rowe SM, Jain R; VX17-445-102 Study Group. Elexacaftor-Tezacaftor-Ivacaftor for Cystic Fibrosis with a Single Phe508del Allele. N Engl J Med. 2019 Nov 7;381(19):1809-1819. doi: 10.1056/NEJMoa1908639. Epub 2019 Oct 31. PMID 31697873
- [Background] Gifford AH, Mayer-Hamblett N, Pearson K, Nichols DP. Answering the call to address cystic fibrosis treatment burden in the era of highly effective CFTR modulator therapy. J Cyst Fibros. 2020 Sep;19(5):762-767. doi: 10.1016/j.jcf.2019.11.007. Epub 2019 Nov 21. PMID 31761739
- [Background] Donaldson SH, Laube BL, Corcoran TE, Bhambhvani P, Zeman K, Ceppe A, Zeitlin PL, Mogayzel PJ Jr, Boyle M, Locke LW, Myerburg MM, Pilewski JM, Flanagan B, Rowe SM, Bennett WD. Effect of ivacaftor on mucociliary clearance and clinical outcomes in cystic fibrosis patients with G551D-CFTR. JCI Insight. 2018 Dec 20;3(24):e122695. doi: 10.1172/jci.insight.122695. PMID 30568035
- [Background] Klijn PH, van Stel HF, Quittner AL, van der Net J, Doeleman W, van der Schans CP, van der Ent CK. Validation of the Dutch cystic fibrosis questionnaire (CFQ) in adolescents and adults. J Cyst Fibros. 2004 Mar;3(1):29-36. doi: 10.1016/j.jcf.2003.12.006. PMID 15463884